CLINICAL TRIAL: NCT05031845
Title: Identification of Potentially Long-term Pulmonary Complications of COVID-19: A Pilot Study of Low-Dose Chest CT (LDCT) Imaging
Brief Title: Low-Dose Chest CT (LDCT) COVID-19 Study
Status: Completed | Type: Observational
Sponsor: Kaiser Permanente (Other)
Collaborators: Garfield Memorial Fund (Other)
Responsible Party: Principal Investigator, Douglas W. Roblin, Senior Research Scientists, Kaiser Permanente
Other Study IDs: 1689022
Record Dates: First submitted 2021-08-28; First posted 2021-09-02 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVID-19 positive, Hospitalized with ARDS: 1. Patients with chest imaging at the time of the first COVID-positive PCR test will have their first LDCT within 3 to 4 months after COVID 19 diagnosis. A second LDCT between 3 to 6 months after the initial LDCT.
  2. Patients without chest imaging at the time of the first COVID-positive PCR test or with a negative COVID PCR test will have their first LDCT within 2 weeks to 1 month after their recovery from COVID 19, or testing. A second LDCT may be performed between 3 to 6 months after the initial LDCT.
- COVID-19 positive, not hospitalized with ARDS: 1. Patients with chest imaging at the time of the first COVID-positive PCR test will have their first LDCT within 3 to 4 months after COVID 19 diagnosis. A second LDCT between 3 to 6 months after the initial LDCT.
  2. Patients without chest imaging at the time of the first COVID-positive PCR test or with a negative COVID PCR test will have their first LDCT within 2 weeks to 1 month after their recovery from COVID 19, or testing. A second LDCT may be performed between 3 to 6 months after the initial LDCT.
- COVID-19 negative, not hospitalized with ARDS: 1. Patients with chest imaging at the time of the first COVID-positive PCR test will have their first LDCT within 3 to 4 months after COVID 19 diagnosis. A second LDCT between 3 to 6 months after the initial LDCT.
  2. Patients without chest imaging at the time of the first COVID-positive PCR test or with a negative COVID PCR test will have their first LDCT within 2 weeks to 1 month after their recovery from COVID 19, or testing. A second LDCT may be performed between 3 to 6 months after the initial LDCT.

SUMMARY:
The goal of our proposed pilot study is to collect low dose CT (LDCT) findings from chest evaluations of a representative sample of 120 symptomatic Caucasian and African American, and Hispanic adults (45 each), stratified by presence of acute respiratory distress syndrome (ARDS) and COVID-19 positivity or negative PCR screening results. These data will provide us with preliminary data on the type and extent of alveolar remodeling by race and by severity of recent infectious respiratory disease. Findings from our study would will help us to determine if a larger multi-site research application to NHLBI or a similar funding agency might be possible and provide critical preliminary data on variation in LDCT findings by COVID-19 attributable respiratory health, race, and other risk factors (e.g., smoking history, comorbidities, and socioeconomic status).

DETAILED DESCRIPTION:
This is a prospective data collection study of random samples of Caucasian and African American, and Hispanic adults, who are symptomatic and recently tested with a nasal or nasopharyngeal swab test (PCR test) and by test positivity and/or evidence of recent acute respiratory distress.

Our study has 2 objectives: 1) demonstrate the feasibility of using KP electronic health records (EHR) and associated computerized data resources to identify and recruit representative samples of Caucasian and African American, and Hispanic adults with varying likelihoods of lung remodeling, and 2) identify the implementation opportunities and challenges associated with recruitment for and collection of primary LDCT findings in a representative sample of adults from a diverse urban population.

The specific aims of our study are:

Aim 1: Implement a sampling and recruitment protocol to collect representative samples of Caucasian and African American, and Hispanic adults by clinical history attributable to ARDS (e.g., hospitalization for ARDS, not hospitalized by positive/negative for COVID-19) and presenting with symptoms typical of COVID-19 (i.e. fever, cough, shortness of breath, nausea/vomiting) Aim 2: Collect LDCT findings and self-reported respiratory health at the time of LDCT from this sample.

Aim 3: Link the LDCT findings to other electronic health record (EHR) data to assess face validity of findings through associations with race, other patient demographics, and clinical risk factors associated with self-reported respiratory health.

ELIGIBILITY:
Inclusion Criteria:

* KPMAS members, primarily residing in the DCSM service area (Montgomery, Frederick or Prince George's counties),
* ≥ 18 years of age or older
* Have a recent PCR test with a positive or negative result, and/or evidence of ARDS and who were symptomatic for COVID-19 related symptoms at the time of the test.

Exclusion Criteria:

* Pregnant or intending to become pregnant in the next 1-3 months
* Cancer or other treatment involving radiation therapy at any time
* Terminally ill
* Non-English speaking
* Diminished cognitive capacity
* Developmental disabilities

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eligible participants must be ≥ 18 years of age, alive, and a KPMAS member primarily residing in the DCSM service area (Montgomery, Frederick or Prince George's counties), at the time of invitation and had COVID-19 related symptoms at the time of COVID-19 PCR testing.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
St. George's Respiratory Questionnaire (SGRQ) | Baseline
  The SGRQ is a disease specific quality of life assessment tool validated in both COPD and asthma 12-14. The questionnaire consists of 50 items divided into three parts measuring symptoms, activity limitation and social and emotional impact of disease. The questionnaire will be used to examine respiratory health.
LDCT Abstract Form | Baseline
  LDCT findings will be classified on the presence/absence of ground glass opacities, consolidation, septal thickening, and crazy paving. In addition, the findings will be classified using two quantitative measures: number of lobes involved and percentage of involvement per lobe.
Change from Baseline St. George's Respiratory Questionnaire (SGRQ) | 3 to 6 months after the initial LDCT
  The SGRQ is a disease specific quality of life assessment tool validated in both COPD and asthma 12-14. The questionnaire consists of 50 items divided into three parts measuring symptoms, activity limitation and social and emotional impact of disease. The questionnaire will be used to examine respiratory health.
Change from Baseline LDCT Abstract Form | 3 to 6 months after the initial LDCT
  LDCT findings will be classified on the presence/absence of ground glass opacities, consolidation, septal thickening, and crazy paving. In addition, the findings will be classified using two quantitative measures: number of lobes involved and percentage of involvement per lobe.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas W Roblin, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Mid-Atlantic States Mid-Atlantic Permanente Research Institute, Rockville, Maryland, United States